CLINICAL TRIAL: NCT02360995
Title: The Clinical Investigation of Colgate Total Toothpaste as Compared to Crest Pro-Health Toothpaste and Crest Pro-Health Mouthwash, and Crest Cavity Protection Toothpaste and Crest Fluoride Mouthwash in Reducing Plaque and Gingivitis: A Six-week Clinical Study in the US
Brief Title: The Clinical Investigation of Toothpaste as Compared to Toothpaste and Mouthwash in Reducing Plaque and Gingivitis: A Six-week Clinical Study in the US
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2014-06-PLAGIN-CT-YPZ
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Results first posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2014-05

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Triclosan; hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Total Toothpaste (Active Comparator): Triclosan/fluoride toothpaste
  Interventions: Drug: Triclosan/fluoride toothpaste
- Toothpaste + Mouthwash (Active Comparator): Stannous fluoride toothpaste & cetylpyridinium chloride Mouthwash
  Interventions: Drug: stannous fluoride toothpaste; Drug: cetylpyridinium chloride Mouthwash
- Control group (Placebo Comparator): fluoride toothpaste +fluoride mouthwash
  Interventions: Drug: fluoride toothpaste; Drug: Fluoride Mouthwash

INTERVENTIONS:
Drug: Triclosan/fluoride toothpaste — Brush whole mouth with Total toothpaste (sold in the US), using a Total 360 toothbrush, 2 times/day for 6 weeks (study duration).
  Other Names: Total toothpaste
  Arms: Total Toothpaste
Drug: stannous fluoride toothpaste — Brush whole mouth with Crest Pro-Health toothpaste using an Oral B Pro-Health toothbrush for 1 minute, 2 times/day for 6 weeks (study duration).
  Other Names: Crest Pro-Health toothpaste
  Arms: Toothpaste + Mouthwash
Drug: fluoride toothpaste — Brush whole mouth with Crest Cavity Protection toothpaste using an Oral B Indicator toothbrush for 1 minute, 2 times/day for 6 weeks (study duration).
  Other Names: Crest Cavity Protection toothpaste
  Arms: Control group
Drug: Fluoride Mouthwash — Immediately after each toothbrushing rinse whole mouth with 20 ml of Crest fluoride Mouthrinse for 30 seconds each time.
  Other Names: Crest Pro-Health For Me Breezy Mint mouthwash
  Arms: Control group
Drug: cetylpyridinium chloride Mouthwash — Immediately after each toothbrushing rinse whole mouth with 20 ml of Crest Pro-Health Mouthrinse for 30 seconds each time.
  Other Names: Crest Pro-Health Multi-Protection mouthwash
  Arms: Toothpaste + Mouthwash

SUMMARY:
The objective of this clinical research study is to evaluate clinical efficacy of Colgate Total Toothpaste as compared to Crest Pro-Health Toothpaste and Crest Pro-Health Mouthwash, and Crest Cavity Protection Toothpaste and Crest Fluoride Mouthwash in reducing gingivitis and dental plaque in adults in a six-week clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, ages 18-70, inclusive.
2. Availability for the six-week duration of the clinical research study.
3. Good general health.
4. Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
5. Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
6. Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
7. Signed Informed Consent Form

Exclusion Criteria:

1. Presence of orthodontic bands.
2. Presence of partial removable dentures.
3. Tumor(s) of the soft or hard tissues of the oral cavity.
4. Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
5. Five or more carious lesions requiring immediate restorative treatment.
6. Antibiotic use any time during the one month prior to entry into the study.
7. Participation in any other clinical study or test panel within the one month prior to entry into the study.
8. Dental prophylaxis during the past two weeks prior to baseline examinations.
9. History of allergies to oral care/personal care consumer products or their ingredients.
10. On any prescription medicines that might interfere with the study outcome.
11. An existing medical condition which prohibits eating or drinking for periods up to 4 hours.
12. History of alcohol or drug abuse.
13. Pregnant or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yimimg Li, DDS, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment is completed locally by the clinical site
Pre-assignment Details: There is no wash out or pre-assignment of any study product.
Groups:
- Toothpaste + Mouthwash: Stannous fluoride toothpaste & cetylpyridinium chloride Mouthwash
  stannous fluoride toothpaste & cetylpyridinium chloride Mouthwash: Brush whole mouth with Crest Pro-Health toothpaste using an Oral B Pro-Health toothbrush for 1 minute, 2 times/day for 6 weeks (study duration). Immediately after each toothbrushing rinse whole mouth with 20 ml of Crest Pro-Health Mouthrinse for 30 seconds each time.
- Control Group: fluoride toothpaste +fluoride mouthwash
  fluoride toothpaste + fluoride mouthwash: Brush whole mouth with Crest Cavity Protection toothpaste using an Oral B Indicator toothbrush for 1 minute, 2 times/day for 6 weeks (study duration). Immediately after each toothbrushing rinse whole mouth with 20 ml of Crest fluoride Mouthrinse for 30 seconds each time.
Period: Overall Study
Arm/Group | Total Toothpaste | Toothpaste + Mouthwash | Control Group
Started | 43 | 43 | 43
Completed | 41 | 42 | 41
Not Completed | 2 | 1 | 2
Not completed — Lost to Follow-up | 2 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Toothpaste | Toothpaste + Mouthwash | Control Group | Total
Number analyzed (Participants) | 43 | 43 | 43 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.68 (16.85) | 44.90 (15.51) | 44.39 (13.68) | 44.47 (15.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 24 | 72
  Male | 20 | 18 | 19 | 57
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 43 | 129

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque Scores
Description: Dental Plaque (Quigley-Hein, Turesky Modification Index) Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Toothpaste | Toothpaste + Mouthwash | Control Group
Number analyzed (Participants) | 43 | 43 | 43
units on a scale | 3.91 (0.31) | 3.86 (0.45) | 3.84 (0.23)
Statistical Analysis 1: Comparison: Total Toothpaste vs Toothpaste + Mouthwash vs Control Group; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.652, ANOVA

2. Primary Outcome: Dental Plaque Scores
Description: as for outcome 1
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Total Toothpaste | Toothpaste + Mouthwash | Control Group
Number analyzed (Participants) | 41 | 42 | 41
units on a scale | 3.42 (0.06) | 3.69 (0.06) | 3.73 (0.06)
Statistical Analysis 1: Comparison: Total Toothpaste vs Toothpaste + Mouthwash vs Control Group; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Primary Outcome: Dental Plaque Scores
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Total Toothpaste | Toothpaste + Mouthwash | Control Group
Number analyzed (Participants) | 41 | 42 | 41
units on a scale | 1.05 (0.04) | 1.15 (0.04) | 1.24 (0.04)
Statistical Analysis 1: Comparison: Total Toothpaste vs Toothpaste + Mouthwash vs Control Group; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Primary Outcome: Gingivitis Scores
Description: Gingivitis scale (Loe & Silness Gingival Index) Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Toothpaste | Toothpaste + Mouthwash | Control Group
Number analyzed (Participants) | 43 | 43 | 43
units on a scale | 1.38 (0.22) | 1.35 (0.24) | 1.41 (0.24)
Statistical Analysis 1: Comparison: Total Toothpaste vs Toothpaste + Mouthwash vs Control Group; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.533, ANOVA

5. Primary Outcome: Gingivitis Scores
Description: as for outcome 4
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Total Toothpaste | Toothpaste + Mouthwash | Control Group
Number analyzed (Participants) | 41 | 42 | 41
units on a scale | 1.15 (0.04) | 1.20 (0.04) | 1.30 (0.04)
Statistical Analysis 1: Comparison: Total Toothpaste vs Toothpaste + Mouthwash vs Control Group; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Primary Outcome: Gingivitis Scores
Description: as for outcome 4
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Total Toothpaste | Toothpaste + Mouthwash | Control Group
Number analyzed (Participants) | 41 | 42 | 41
units on a scale | 1.05 (0.04) | 1.15 (0.04) | 1.24 (0.04)
Statistical Analysis 1: Comparison: Total Toothpaste vs Control Group; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline, 4 and 6 weeks
Arm/Group | Total Toothpaste | Toothpaste + Mouthwash | Control Group
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days